CLINICAL TRIAL: NCT05034718
Title: Implementation of the Pittsburgh Infant Brain Injury Score
Acronym: PIBIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: The Beckwith Institute (Other)
Responsible Party: Principal Investigator, Rachel Berger MD, MPH, Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY21010197
Record Dates: First submitted 2021-07-29; First posted 2021-09-05 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Brain Injury; Clinical Decision Support; Infant
MeSH Terms: conditions — Brain Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Completion of nurse powerform and data collection only.
  Interventions: Other: Standard of care
- Intervention Arm (Experimental): Completion of nurse powerform, data collection and physician alert/powerform with score calculation and recommendations.
  Interventions: Other: PIBIS clinical decision support

INTERVENTIONS:
Other: PIBIS clinical decision support — The intervention is the presence of the PIBIS physician alert and powerform, which is clinical decision support for the treating provider if a patient meets inclusion criteria for Pittsburgh Infant Brain Injury Score (PIBIS) calculation.
  Arms: Intervention Arm
Other: Standard of care — Standard of care, absent the PIBIS powerform and alert for providers.
  Arms: Control Arm

SUMMARY:
This is an implementation study of the Pittsburgh Infant Brain Injury Score (PIBIS) into the UPMC Children's Hospital of Pittsburgh emergency department. Children less than 1 year of age presenting to the CHP ED for symptoms which place them at increased risk for AHT as defined in the PIBIS validation study will be potentially eligible.

DETAILED DESCRIPTION:
Abusive head trauma is the leading cause of death due to physical abuse. Missing the diagnosis of abusive head trauma (AHT), particularly when it less severe is common and contributes to increased morbidity and mortality. Over the past 10 years, the investigators have derived and subsequently prospectively validated the Pittsburgh Infant Brain Injury Score (PIBIS), a point of care clinical decision rule to help physicians determine when it is appropriate to obtain neuroimaging in infants who present to the ED for evaluation of soft neurologic signs such as vomiting and fussiness. The results of the NIH multi-center prospective validation were published in 2016 in Pediatrics.

The next step in evaluating PIBIS as a clinical prediction rule is to perform an implementation study. Children less than 1 year of age presenting to the CHP ED for symptoms which place them at increased risk for AHT as defined in the PIBIS validation study will be potentially eligible.

Discrete fields in the electronic health record - including patient age, Emergency Severity Index (ESI), Glasgow Coma Scale (GCS) score, temperature and chief complaint - will be used to identify potentially eligible children in a systematic and efficient manner. Children who are potentially eligible based on this initial screen will trigger an alert to the nurse who will then complete a brief powerform to ensure eligibility and assess for inclusion/exclusion criteria. Due to the nature of the research, the investigators will seek a waiver of informed consent as has been done in similar studies at our institution and others. At this point, eligible children will be considered enrolled.

For children enrolled during the intervention period, providers will be presented with a detailed decision support strategy which encourages - but does not require - use of the PIBIS to make clinical decision re: the need for neuroimaging. For children enrolled during the control period, no other clinical decision support will occur. The duration of this evaluation period will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 days to less than 1 year
* Chief complaint of Apnea, BRUE, Fussiness or Irritability, Lethargy, Neurologic complaint, Poor Feeding-Acute, Seizures/Spells, or Vomiting Alone
* First temperature in the ED less than or equal to 38.3C
* Acuity level/ESI of 3, 4, or 5

Exclusion Criteria:

* History of trauma related to this ED encounter
* Parent reported temperature of greater than 38.3C in the prior 24 hours
* Prior abnormal neuroimaging
* Previously enrolled in this study within preceding 28 days
* Provider preference for any reason

Ages: 30 Days to 364 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1989 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Eligibility confirmation | From enrollment to hospital discharge, up to one month
  Children identified as eligible by Cerner and confirmed by the nurse powerform as eligible for PIBIS will also be determined to be eligible after chart review and discussion with the clinician (which is how eligibility was determined during the validation study). The primary outcome will be the concordance between these two methods of determining eligibility. A concordance of >90% is the goal.
Proportion of children with PIBIS calculation and recommendations | From enrollment to hospital discharge, up to one month
  The proportion of children eligible for PIBIS who
  1. have a PIBIS score calculated and
  2. in whom the provider follows the recommendation by PIBIS OR documents in the EHR the clinical reasoning why they are NOT following the recommendation (e.g. patient being admitted, in-patient team will make decision).

SECONDARY OUTCOMES:
Proportion of children who undergo neuroimaging (head CT or brain MRI) during the control and intervention periods | From enrollment to hospital discharge, up to one month
  The proportion of children eligible for PIBIS who undergo neuroimaging (head CT or brain MRI) during the control and intervention periods
Proportion of neuroimaging which demonstrates an abnormality during the control and intervention periods | From enrollment to hospital discharge, up to one month
  Proportion of neuroimaging which demonstrates an abnormality during the control and intervention periods
Proportion of all children with each PIBIS score who are ultimately diagnosed with physical abuse by the CHP Child Protection Team | From enrollment to hospital discharge, up to one month
  Proportion of all children with each PIBIS score who are ultimately diagnosed with physical abuse by the CHP Child Protection Team
The number of enrolled children who return to the ED within 6 months of enrollment and undergo neuroimaging. | From enrollment to 6 months following hospital discharge
  The number of enrolled children who return to the ED within 6 months of enrollment and undergo neuroimaging.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Berger, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No